CLINICAL TRIAL: NCT02798835
Title: Adductor Canal Block: Single Injection vs Catheter for Pain Management of Total Knee Arthroplasty - A Randomized, Unblinded, Non-Inferiority Trial
Brief Title: Single Injection Adductor Canal Block vs Catheter for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Steven Lee, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-01058
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Dexamethasone; Bupivacaine; Fentanyl; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adductor Canal block (Active Comparator): Postoperatively in the PACU, this group will receive 20ml 0.5% ropivacaine for their ACB.
  Interventions: Drug: Adductor canal block; Drug: Bupivacaine; Drug: Fentanyl; Drug: Ropivacaine 0.5% Injectable Solution
- Adductor canal block with dexamethasone (Active Comparator): Postoperatively in the PACU, this group will receive 20ml 0.5% ropivacaine for their ACB along with 8mg IV dexamethasone.
  Interventions: Drug: Adductor canal block with dexamethasone; Drug: Bupivacaine; Drug: Fentanyl; Drug: Ropivacaine 0.5% Injectable Solution; Drug: Dexamethasone
- Adductor canal catheter (Active Comparator): Postoperatively in the PACU, this group will receive 20ml 0.5% ropivacaine for their adductor canal block and have a catheter placed in the adductor canal at the mid-thigh. 0.2% ropivacaine at 5ml/hr will be run for 48 hours.
  Interventions: Drug: Adductor canal catheter; Drug: Bupivacaine; Drug: Fentanyl; Drug: Ropivacaine 0.5% Injectable Solution

INTERVENTIONS:
Drug: Adductor canal block — Spinal anesthesia with 2-3 ml 0.5% bupivacaine and 0-20mcg of fentanyl. At the end of the case, the surgeon will infiltrate 30ml 0.5% ropivacaine peri-articularly. 20ml 0.5% ropivacaine in the adductor canal in PACU.
  Arms: Adductor Canal block
Drug: Adductor canal block with dexamethasone — Spinal anesthesia with 2-3 ml 0.5% bupivacaine and 0-20mcg of fentanyl. At the end of the case, the surgeon will infiltrate 30ml 0.5% ropivacaine peri-articularly. 20ml 0.5% ropivacaine in the adductor canal along with 8mg dexamethasone IV in PACU.
  Arms: Adductor canal block with dexamethasone
Drug: Adductor canal catheter — Spinal anesthesia with 2-3 ml 0.5% bupivacaine and 0-20mcg of fentanyl. At the end of the case, the surgeon will infiltrate 30ml 0.5% ropivacaine peri-articularly. 20ml 0.5% ropivacaine and a catheter placed in PACU, with a continuous infusion of 0.2% ropivacaine started.
  Arms: Adductor canal catheter
Drug: Bupivacaine — Used in spinal anesthetic
Drug: Fentanyl — May or may not be used in spinal anesthetic
Drug: Ropivacaine 0.5% Injectable Solution — Local anesthetic to be used by surgeon as local infiltration and by anesthesiologist in adductor canal block.
Drug: Dexamethasone — To be given intravenously at time of nerve block to one of the study arms.
  Arms: Adductor canal block with dexamethasone

SUMMARY:
This study investigates single injection adductor canal block (ACB) with or without intravenous dexamethasone and adductor canal catheter for pain management of total knee arthroplasty. This is a non-inferiority trial seeking to determine whether single injection ACB with dexamethasone is "no worse" than a continuous catheter.

DETAILED DESCRIPTION:
1. Purpose

   To determine whether single shot adductor canal nerve blocks with intravenous dexamethasone are non-inferior to continuous adductor canal blockade.
2. Hypotheses

   The use of adductor canal nerve block with intravenous dexamethasone will not be inferior to continuous adductor canal blockade for opioid requirements 24h post operatively.

   The single injection adductor canal block without dexamethasone will have the most opioid consumption. The dexamethasone and catheter groups will be superior to single injection alone in terms of 12 and 48h opioid consumption, length of stay, anti-emetic usage, pain score and quality of recovery score.
3. Justification

   Total knee arthroplasty is a very commonly performed operation in North America, with a high propensity for postoperative pain. Inadequate analgesia limits functional recovery and leads to delays in hospital discharge, as a result of poor mobility. Effective analgesia allows for earlier mobilization and improved postoperative recovery, with a multi-modal regime being the ideal method to achieve this.

   Currently a multi-modal regime is provided to patients: intraoperatively with a neuraxial technique (spinal anesthesia), along with surgeon infiltrated local anesthetic at the end of the operation, and then postoperatively using systemic opioids via patient controlled analgesia (PCA). Opioids have many side effects, including nausea and vomiting, sedation, respiratory depression and urinary retention. These all lead to delay in ambulation and recovery.

   Many centers now incorporate peripheral nerve blocks as part of the multi-modal analgesic regime, with continuous femoral nerve blockade being commonly used for analgesia. This does decrease the amount of postoperative opioid used, but has the downside of causing quadriceps muscle weakness leading to an increased risk of falls and delayed ambulation. For this reason, there has been an increase in the use of the adductor canal block, a nerve block of the distal femoral nerve at the mid-thigh level, that has been shown to preserve quadriceps function better than a femoral nerve block, whilst still ensuring decreased opioid use. To date, no studies have compared single shot adductor canal block with continuous adductor canal blockade, but both have been shown to be comparable to femoral nerve blockade, whilst decreasing the likelihood of quadriceps muscle weakness.

   Further to this, it has been shown that the addition of dexamethasone, administered via the intravenous or perineural route to peripheral nerve blockade, prolongs the duration of analgesia. Perineural administration of dexamethasone is an off label use and there is also a theoretical risk of neurotoxicity from dexamethasone itself. Findings to date indicate that the efficacy of dexamethasone administered intravenously is non-inferior to perineural injection. Both routes prolong the analgesic benefit of peripheral nerve blocks with similar reductions in opioid requirements.

   Opioid PCA is the most commonly used modality for postoperative analgesia following total knee arthroplasty. The information from this study will enable ascertainment of the best method for allowing patients good functional recovery, whilst minimizing opioid side effects.
4. Objectives

   The primary aim of this study is to compare the efficacy of adductor canal nerve block, with and without intravenous dexamethasone, and continuous adductor canal blockade with a catheter to ascertain cumulative opioid consumption post-operatively. Specifically, the trial seeks to answer whether the adductor canal block with dexamethasone fares no worse (non-inferior) than a continuous catheter.

   The secondary aims are to compare the quality of anesthesia recovery using the QoR-40 questionnaire administered at 48 hours postoperatively, pain score, length of hospital stay, complications of nerve blockade, incidence of catheter dislodgement and opioid side effects (nausea/vomiting) with the different techniques.
5. Research Methods

   Trial Design

   This will be a randomize controlled, non-blinded, non-inferiority trial, involving patients having primary unilateral total knee arthroplasty. There are three arms: adductor canal single injection (baseline control), adductor canal single injection plus dexamethasone (test intervention) and adductor canal catheter (active control).

   Setting

   This will be a single-centre trial at UBC Hospital (UBCH).

   B. Randomization

   Prior to surgery, for each consented patient, a sealed unmarked opaque envelope will be opened to determine the modality of analgesia that the patient will receive. The patients will either receive an adductor canal block postoperatively, an adductor canal block postoperatively along with intravenous dexamethasone, or have an adductor canal catheter placed postoperatively for continuous adductor canal blockade.

   D. Data Collection

   Demographic data including patient age, sex, height, weight, BMI, and medications including analgesics, comorbidities and American Society of Anesthesia (ASA) classification will be determined from the anesthetic record.

   Numerical Rating Scale (NRS) pain scores from 0-10 as well as cumulative opioid consumption in oral morphine equivalents will be determined at set time points of 12, 24, 48 hours. The data will be determined from the patient's pain flow sheet and medication administration record (MAR), which are part of the standard charting found on the hospital ward. Opioid data from PCA will be obtained from the hospital database which electronically logs usage. The patient's chart will also be used to note anti-emetic medication usage. At 48 hours, all participants will be provided with a QoR-40 questionnaire, a validated 40 item questionnaire on the quality of recovery from anesthesia. The time of discharge will be recorded from the hospital data base.

   Complications from adductor canal catheters will be recorded, such as catheter dislodgement and site infection. For patients unable to complete the study, the reason will be noted and data will be included in an intention to treat analysis.

   E. Statistical Analysis

   Sample Size:

   The investigators do not have institutional data of standard deviation (SD) of morphine equivalent consumption for primary total knee arthroplasty. Based on previous studies, the standard deviation of morphine equivalent consumption at 24h is estimated to be 20 mg IV. We consider a reduction of 10 mg to be clinically relevant at this time point and therefore set it as the non-inferiority margin. Using the following online calculator: https://www.sealedenvelope.com/power/continuous-noninferior/ based on a power of 80% and significance level of 5%, the number of patients required per group is 50. The aim is to recruit 60 patients per group to account for potential drop outs.
6. Data Analysis: Categorical data will be analysed with chi-squared tests. Numeric variables will be compared with independent T-tests if distributions were normal. If Kolmogorov-Smirnoff test for normality of distribution was significant non-parametric Mann Whitney U tests will be utilized. Statistical significance will be assumed if P <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients over or equal to the age of 18 years old who can understand the study protocol and are able to give consent
* Patients with an American Society of Anaesthesiology (ASA) classification 1 to 3
* Patients must have a preoperative oral 24 hour opioid consumption of less than or equal to 30 mg morphine equivalents
* Patients must be able to understand and be able to use patient controlled analgesia
* Patients must be undergoing a primary total knee arthroplasty with neuraxial anesthesia

Exclusion Criteria:

* Patients with a contraindication to neuraxial and/or regional anaesthesia
* Patients with an allergy to local anaesthetics
* Patients who have chronic pain not related to their knee joint
* Patients with chronic opioid use (daily or almost daily use >3 months)
* Patients with contraindications to dexamethasone (allergy, infection, Insulin dependent Diabetes Mellitus)
* Patients with pre-existing neuropathy
* Patients with hepatic failure
* Patients with renal failure with eGFR<60
* Patients with allergy to ketorolac or NSAIDs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lee, MD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perlas A, Kirkham KR, Billing R, Tse C, Brull R, Gandhi R, Chan VW. The impact of analgesic modality on early ambulation following total knee arthroplasty. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):334-9. doi: 10.1097/AAP.0b013e318296b6a0. PMID 23759708
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Allen HW, Liu SS, Ware PD, Nairn CS, Owens BD. Peripheral nerve blocks improve analgesia after total knee replacement surgery. Anesth Analg. 1998 Jul;87(1):93-7. doi: 10.1097/00000539-199807000-00020. PMID 9661553
- [Background] Charous MT, Madison SJ, Suresh PJ, Sandhu NS, Loland VJ, Mariano ER, Donohue MC, Dutton PH, Ferguson EJ, Ilfeld BM. Continuous femoral nerve blocks: varying local anesthetic delivery method (bolus versus basal) to minimize quadriceps motor block while maintaining sensory block. Anesthesiology. 2011 Oct;115(4):774-81. doi: 10.1097/ALN.0b013e3182124dc6. PMID 21394001
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Abdallah FW, Johnson J, Chan V, Murgatroyd H, Ghafari M, Ami N, Jin R, Brull R. Intravenous dexamethasone and perineural dexamethasone similarly prolong the duration of analgesia after supraclavicular brachial plexus block: a randomized, triple-arm, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):125-32. doi: 10.1097/AAP.0000000000000210. PMID 25629321
- [Background] Rahangdale R, Kendall MC, McCarthy RJ, Tureanu L, Doty R Jr, Weingart A, De Oliveira GS Jr. The effects of perineural versus intravenous dexamethasone on sciatic nerve blockade outcomes: a randomized, double-blind, placebo-controlled study. Anesth Analg. 2014 May;118(5):1113-9. doi: 10.1213/ANE.0000000000000137. PMID 24686045
- [Derived] Lee S, Rooban N, Vaghadia H, Sawka AN, Tang R. A Randomized Non-Inferiority Trial of Adductor Canal Block for Analgesia After Total Knee Arthroplasty: Single Injection Versus Catheter Technique. J Arthroplasty. 2018 Apr;33(4):1045-1051. doi: 10.1016/j.arth.2017.11.018. Epub 2017 Nov 16. PMID 29198872

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Started | 60 | 60 | 60
Completed | 60 | 60 | 57
Not Completed | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter | Total
Number analyzed (Participants) | 60 | 60 | 57 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8.9) | 64.6 (9.1) | 65.6 (7.7) | NA (NA)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 42 | 33 | 112
  Male | 23 | 18 | 24 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (5.8) | 29.6 (6.1) | 29.9 (5) | NA (NA)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative 24 Hour Oral Morphine Equivalent Consumption
Description: Post-operative analgesia at 24 hours
Time Frame: 24 hours (Day 1)
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
mg | 111.8 [79.5 to 150] | 118 [69 to 155.8] | 153 [100.5 to 170]

2. Secondary Outcome: Cumulative 12 Hour Oral Morphine Equivalent Consumption
Description: Post-operative analgesia at 12 hours
Time Frame: 12 hours (Day 0)
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
mg | 61.5 [40.8 to 75] | 49.5 [30 to 82.5] | 82 [49 to 104]

3. Secondary Outcome: Cumulative 48 Hour Oral Morphine Equivalent Consumption
Description: Post-operative analgesia at 48 hours
Time Frame: 48 hours (Day 2)
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
mg | 192.9 [137.6 to 274] | 196 [127.9 to 277.5] | 223.5 [175.5 to 282]

4. Secondary Outcome: Pain Score
Description: Patient's level of pain using NRS (Numeric Ratings Scale) pain scale where the range is 0 (no pain) to 10 (worst pain)
Time Frame: 12, 24 and 48 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
score on a scale
  12h | 3 [2 to 4] | 3 [2 to 4] | 4 [3 to 4]
  24h | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
  48h | 2 [2 to 3] | 3 [2 to 4] | 3 [2 to 4]

5. Secondary Outcome: Quality of Recovery (QoR-40)
Description: Quality of recovery measured using the QoR-40 at 48 hours postoperatively. This is a validated scale where a higher score denotes better recovery/satisfaction after surgery. The range is 40-200.
Time Frame: 48 hours (Day 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
score on a scale | 160.5 (20.1) | 166.5 (19.3) | 167.2 (17.5)

6. Secondary Outcome: Length of Stay
Description: Time to hospital discharge
Time Frame: From surgical date until hospital discharge, up to 3 weeks
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
hours | 70.8 [66.9 to 96.5] | 71.5 [66.3 to 89.3] | 71.5 [65.8 to 94.3]

7. Secondary Outcome: Incidence of Participants With Nausea/Vomiting Requiring Anti-emetics
Description: Number of Participants with Nausea/Vomiting requiring anti-emetics from 0-48 hours after surgery.
Time Frame: 0 to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
Participants
  0-12h | 19 | 14 | 19
  12-24h | 26 | 17 | 24
  24-48h | 15 | 17 | 17

8. Secondary Outcome: Time to First Use of PCA
Description: from time zero to first press of PCA button
Time Frame: 0 to 48 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
hours | 4.1 [2.6 to 5.1] | 4.9 [3.4 to 6.1] | 3.8 [3 to 5]

9. Other Pre Specified Outcome: Adductor Canal Block Complications
Description: Incidence of catheter dislodgement or site infection
Time Frame: From time of catheter insertion until catheter removal, up to Day2/48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
Participants | 0 | 0 | 0

10. Other Pre Specified Outcome: Nerve Block Complications
Description: Nerve block complications at any time point during study
Time Frame: 0 to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
Number analyzed (Participants) | 60 | 60 | 57
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From surgery completion to time of discharge
Arm/Group | Adductor Canal Block | Adductor Canal Block With Dexamethasone | Adductor Canal Catheter
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/57
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No